CLINICAL TRIAL: NCT02023502
Title: Proteomic Pattern in Female Stress Urinary Incontinence: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marianne Koch, Principal Investigator, Medical University of Vienna
Other Study IDs: EK 1788/2013
Record Dates: First submitted 2013-11-18; First posted 2013-12-30 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Female Stress Urinary Incontinence
Keywords: female stress urinary incontinence; proteomics; biomarker
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- stress urinary incontinence: Patients presenting with stress urinary incontinence according to the inclusion and exclusion criteria
  Interventions: Other: collection of urine and blood sample
- healthy controls: healthy women with the same inclusion and exclusion criteria as the case group, except for stress urinary incontinence
  Interventions: Other: collection of urine and blood sample

INTERVENTIONS:
Other: collection of urine and blood sample

SUMMARY:
Objective: The primary objective of the study is the comparison of protein concentrations between patients with stress urinary incontinence (SUI) and healthy controls.

Aim: This pilot study aims to determine a possible altered protein profile in women suffering from SUI, compared to healthy women and therefore to discriminate a potential protein biomarker for SUI.

Main outcome measure: mass spectrometric measuring of urinary proteomic secretome in diseased and healthy subjects (sequence coverage and number of identified proteins)

Trial design: Prospective case- control study

Setting: Department of Gynecology and Obstetrics of the Medical University of Vienna in co- operation with the Core Facilities Proteomics of the Medical University of Vienna

Population: Twenty female patients with SUI and twenty healthy patients who attend the outpatient clinic of the Department of Obstetrics and Gynaecology, Medical University of Vienna (sample size calculation FDR 0.05, power of 80%, assumed proportion of true H0 0.95, assumed standardized effect size of 1)

Methods: Examinations to be carried out: patient history, provocative stress test, ICIQ short form questionnaire, residual urine volume (ultrasound) and urine analysis (dipstick testing). A urine sample is obtained from the patient after spontaneous micturition, to which protease inhibitor will be added immediately. Two serum blood vials (each 9ml) are taken from a peripheral vein of the patient for routine laboratory and further research.

Proteomics analysis will be performed using chromatographic separation (LC) with mass spectrometric detection (MS).

DETAILED DESCRIPTION:
Methods:

Sample preparation and analysis will include:

1. Sample collection and immediate addition of protease inhibitor cocktail (Roche, Complete Protease Inhibitor Cocktail).
2. Urine centrifugation and filtration for removal of cell debris.
3. Protein precipitation by applying methanol/chloroform separation for removal of all possible non-proteinic substances.
4. Protein digestion applying in-solution trypsin, pepsin, and Glu-C.
5. Peptide separation using nano HPLC and different chromatographic approaches.

   1. Reversed phase (RP) separation of peptides and MS detection
   2. Separation of peptides using HILIC (hydrophilic Interaction Liquid Chromatography) for discrimination of polar peptides.
   3. In addition to RP and HILIC directly coupled to MS, digested peptides will be separated using multidimensional approaches. Weak anion exchange columns operated under HILIC conditions will be used to separate peptides carrying posttranslational modifications such as phosphorylation or acetylation, thus, increasing the dynamic range of detection. During this separation, fractions will be collected and re-injected onto the RP and HILIC with MS detection.
   4. All nano HPLC separations will be performed using biocompatible separation system.

Mass spectrometric analysis of digested peptides will be performed using two different detection methods: ion-trap and the time-of-flight (qToF) MS. qToF mass spectrometric detection and analysis will also be used for the label-free quantitation of peptides and proteins detected in samples. All measurements will be performed in triplicate to provide corrections for technical variability of separation and ionization.

General database search will be performed using the Human SwissProt Database in its actual version at the time of analysis. Data search will be performed using Mascot (http://www.matrixscience.com/) and X!Tandem (http://www.thegpm.org/tandem/) search machines, and the final data allocation and filtering by using Scaffold (www.proteomsoftware.com).

Statistical analysis:

Data analysis will be conducted with the bioconductor package limma. Before data analysis, data will be filtered by excluding proteins with measurements with a low interquartile range. Groups will be compared by moderated paired t-statistics adjusting for age. Adjustment for multiple testing will be done by Benjamini-Hochberg correction controlling the FDR at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients with stress urinary incontinence: a history of symptoms of stress urinary incontinence for at least 3 months (including anamnestic complaints of involuntary leakage on effort or exertion or on sneezing or coughing) and a positive provocative stress test (defined as an observed transurethral loss of urine that was simultaneous with a cough or Valsalva maneuver at a bladder volume of 300ml or less)
* patients capable of independent toiling
* patients who are able to fully understand all study procedures and to provide written informed consent to study participation
* age ≥ 18
* patients after vaginal delivery

Exclusion Criteria:

* patients who have previously been treated for SUI (both surgical or pharmacological treatment)
* patients who have a medical history of uncontrolled overactive bladder (OAB) or urinary incontinence other than SUI (including anamnestic complaints on involuntary urine leakage accompanied by or immediately preceded by urgency, not stress induced)
* patients with well established neurological disorder (e.g. Multiple Sclerosis, Parkinson's disease, Alzheimer's disease)
* patients with pelvic organ prolapse stage ≥ II (ICS classification)
* patients with a clinically significant bladder outlet obstruction and/or patients with a post void residual volume (PVR) > 100ml
* patients with a history of acute urinary retention or history of repeated catheterizations due to acute urinary retention within the last 3 months prior to the day of informed consent
* patients with an indwelling catheter and patients practicing intermittent self- catheterization
* patients who have undergone a bladder biopsy or any other minor pelvic surgical intervention less than 30 days prior to the day of informed consent
* patients with a history of bladder cancer
* patients with acute or recurrent urinary tract infection and/or unexplained haematuria
* patients with stone(s) in the bladder or urethra and upper tract stone disease causing symptoms
* patients with evidence of renal insufficiency (creatinine > 1.5x upper limit of normal)
* patients with evidence of hepatic disease (total bilirubin >1.5x upper limit of normal, or AST or ALT or alkaline phosphatase >2x upper limit of normal)
* patients with a history of alcohol and/or other drug abuse
* patients who are unable and/or unlikely to comprehend and follow the study procedures and instructions
* patients who are pregnant or lactating
* patients with serious medical conditions who, in the opinion of the investigators, should not participate in this study

The control group is represented by patients with the same inclusion and exclusion criteria as the case group, except stress urinary incontinence.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the urogynaecology and general gynecology outpatient clinic of the Department of Obstetrics and Gynaecology at the Medical University of Vienna
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
mass spectrometric measuring of urinary proteomic secretome in diseased and healthy subjects (sequence coverage and number of identified proteins) | The primary outcome measure will be assessed for each participant in a time frame of 4-7 days after recruitment
  Comparison of protein concentrations based on number of identified proteins and mass spectrometric spectral count for patients with stress urinary incontinence and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Kölbl, Univ.-Prof.Dr.Dr.h.c., Principal Investigator — Medical University of Vienna, Department of Obstetrics and Gynaecology
Locations (1):
- Medical University of Vienna, Department of Obstetrics and Gynaecology, Vienna, Austria

REFERENCES:
- [Background] Mushkat Y, Bukovsky I, Langer R. Female urinary stress incontinence--does it have familial prevalence? Am J Obstet Gynecol. 1996 Feb;174(2):617-9. doi: 10.1016/s0002-9378(96)70437-4. PMID 8623794
- [Background] Elia G, Bergman J, Dye TD. Familial incidence of urinary incontinence. Am J Obstet Gynecol. 2002 Jul;187(1):53-5. doi: 10.1067/mob.2002.124842. PMID 12114888
- [Background] Chen B, Wen Y, Zhang Z, Guo Y, Warrington JA, Polan ML. Microarray analysis of differentially expressed genes in vaginal tissues from women with stress urinary incontinence compared with asymptomatic women. Hum Reprod. 2006 Jan;21(1):22-9. doi: 10.1093/humrep/dei276. Epub 2005 Aug 26. PMID 16126751
- [Background] Hu S, Loo JA, Wong DT. Human body fluid proteome analysis. Proteomics. 2006 Dec;6(23):6326-53. doi: 10.1002/pmic.200600284. PMID 17083142
- [Background] Ho L, Sharma N, Blackman L, Festa E, Reddy G, Pasinetti GM. From proteomics to biomarker discovery in Alzheimer's disease. Brain Res Brain Res Rev. 2005 Apr;48(2):360-9. doi: 10.1016/j.brainresrev.2004.12.025. PMID 15850675
- [Background] Semmes OJ, Feng Z, Adam BL, Banez LL, Bigbee WL, Campos D, Cazares LH, Chan DW, Grizzle WE, Izbicka E, Kagan J, Malik G, McLerran D, Moul JW, Partin A, Prasanna P, Rosenzweig J, Sokoll LJ, Srivastava S, Srivastava S, Thompson I, Welsh MJ, White N, Winget M, Yasui Y, Zhang Z, Zhu L. Evaluation of serum protein profiling by surface-enhanced laser desorption/ionization time-of-flight mass spectrometry for the detection of prostate cancer: I. Assessment of platform reproducibility. Clin Chem. 2005 Jan;51(1):102-12. doi: 10.1373/clinchem.2004.038950. PMID 15613711
- [Background] Petricoin EF, Ardekani AM, Hitt BA, Levine PJ, Fusaro VA, Steinberg SM, Mills GB, Simone C, Fishman DA, Kohn EC, Liotta LA. Use of proteomic patterns in serum to identify ovarian cancer. Lancet. 2002 Feb 16;359(9306):572-7. doi: 10.1016/S0140-6736(02)07746-2. PMID 11867112